CLINICAL TRIAL: NCT01125332
Title: Evaluation of Topic Anaesthesia for Laryngoscopy With Fibroscopy During Paediatric ENT Consultation
Brief Title: Evaluation of Topic Anaesthesia for Laryngoscopy With Fibroscopy During Paediatric Ear Nose Throat (ENT)Consultation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009 10; 2009-011010-23 (EudraCT Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Nasofibroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group gel KY (Placebo Comparator)
  Interventions: Drug: Indirect laryngoscopy in the flexible nasofibroscope
- group gel lidocaine (Experimental)
  Interventions: Drug: Indirect laryngoscopy in the flexible nasofibroscope

INTERVENTIONS:
Drug: Indirect laryngoscopy in the flexible nasofibroscope
  Arms: group gel KY
Drug: Indirect laryngoscopy in the flexible nasofibroscope
  Arms: group gel lidocaine

SUMMARY:
The purpose of this work is to estimate the efficiency in terms of pain of the application of a local anesthetic (xylocaïne viscous 2%®) during the realization of an examination in naso-fiberscopy in consultation of ENT at the child from 3 to 7 years old.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 4 to 7 years old (old enough to answer the test of self-assessment, the scale of faces)
* Appearing at the consultation of pediatric ENT, requiring an indirect laryngoscopy in the naso-fiberscope for a laryngeal evaluation.
* Subjects girls or boys

Exclusion Criteria:

* All the criteria dissuading the employment of a local anesthetic
* Naso-fibroscopie realized within the framework of a nasal obstruction, or of a balance sheet of the gulp.
* Patients having already been examined by naso-fiberscopy, so that their reactions and their answers are not influenced by the previous experience of the examination.
* Not consent of one of both holders of the parental authority

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
efficacity of local anesthetic
  The purpose of this work is to estimate the efficiency in terms of pain of the application of a local anesthetic (xylocaïne viscous 2%®) during the realization of an examination in naso-fiberscopy in consultation of ENT at the child from 3 to 7 years old.

SECONDARY OUTCOMES:
pain's scale
  The child estimates his(her) own pain by postponing her(it) on a scale of more or less painful faces.

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD NICOLLAS, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assisatnce Publique Hopitaux de Marseille, Marseille, France